CLINICAL TRIAL: NCT03968952
Title: SMARThealth Pregnancy: A Pilot Cluster Randomised Study to Assess Feasibility & Acceptability of a Complex Intervention Using Mobile Decision Support to Detect, Refer & Manage Pregnant Women at High Risk of Future Cardiometabolic Disorders in Rural India.
Brief Title: SMARThealth Pregnancy: Feasibility & Acceptability of a Complex Intervention for High-risk Pregnant Women in Rural India.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: The George Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-19
Record Dates: First submitted 2019-05-23; First posted 2019-05-30 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Pre-Eclampsia; Gestational Diabetes; Anemia
Keywords: Digital health; Gestational Diabetes; Hypertension; Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia; Diabetes, Gestational; Anemia; Hypertension

STUDY DESIGN:
Intervention Model Description: Intervention group cluster will use the SMARThealth Pregnancy training package and mHealth platform. The Control group will have enhanced standard antenatal and postnatal care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMARThealth Pregnancy (Active Comparator): The components of the SMARThealth Pregnancy intervention include:
  1. Educational and Training component on high-risk pregnancy conditions, focusing on; Anaemia, Hypertensive Disorders of Pregnancy (HDPs) and Gestational diabetes mellitus (GDM).
  2. An mHealth platform providing clinical decision support, lifestyle advice, recall and reminder system for Community Health Workers (CHWs) and Primary Care Physicians (PCPs).
  Pregnant women in the intervention group will receive 3 visits at home by their CHW, in addition to their standard antenatal and postnatal care. One visit during the third trimester of pregnancy; one during Week 1 postpartum and; one visit during Week 6 postpartum.
  Interventions: Other: SMARThealth Pregnancy
- Enhanced Standard Care (No Intervention): The control group will receive enhanced standard antenatal and postnatal care, involving:
  1. An awareness programme for pregnant women, Community Health Workers (CHWs) and Primary Care Physicians (PCPs), held at the villages within the control group Primary Health Centre (PHC) cluster (Enhanced Standard Care). The community and health professionals will receive information on the high-risk conditions of anaemia in pregnancy, HDPs and GDM as part of the awareness programme.
  2. Standard antenatal and postnatal care (consisting of free monthly antenatal care, and up to 7 postnatal visits), delivered by CHWs in partnership with their PHC doctor.

INTERVENTIONS:
Other: SMARThealth Pregnancy — Education and Training package on high-risk pregnancies and the associated long-term cardiometabolic risks; An mHealth platform providing mobile decision support to Community Health Workers.
  Arms: SMARThealth Pregnancy

SUMMARY:
Background: Pregnancy-related conditions including hypertensive disorders of pregnancy (HDPs) and gestational diabetes mellitus (GDM) carry independent risks for future cardiovascular disease in women. Early identification, referral and management of pregnant women at increased risk of future cardiometabolic disorders may offer opportunities for prevention.

Objective: To determine the feasibility and acceptability of the SMARThealth Pregnancy intervention to improve the detection, referral and management of pregnant women at high-risk of future cardiometabolic disorders in rural India.

Study design: Cluster randomised pilot study of 4 primary care centres (PHCs) in two diverse areas of rural India.

Outcome: The primary objective of this pilot study is to address the feasibility of the SMARThealth Pregnancy intervention.

DETAILED DESCRIPTION:
Background: Cardiovascular disease (CVD) is the leading cause of death in women in India, and the prevalence of cardiometabolic disorders is rising. Women in rural India (where two-thirds of the population live), are particularly vulnerable due to limited knowledge and healthcare access. Pregnancy-related conditions including hypertensive disorders of pregnancy (HDPs) and gestational diabetes mellitus (GDM) carry independent risks for future cardiovascular disease in women. Early identification, referral and management of pregnant women at increased risk of future cardiometabolic disorders may offer opportunities for prevention. Innovative solutions are required to address the needs of rural women, particularly during the transitions between antenatal and postpartum care and adult health services.

Objective: To determine the feasibility and acceptability of the SMARThealth Pregnancy intervention to improve the detection, referral and management of pregnant women at high-risk of future cardiometabolic disorders in rural India.

Study design: This is a pilot study, using an un-blinded, parallel group, cluster randomised controlled study design.

Study Sites: Jhajjar District, Haryana and Guntur District, Andhra Pradesh, India.

Primary outcome: The primary objective of this pilot study is to address the uncertainties around feasibility: (i) how many PHCs accepted the invitation to participate in a trial; (ii) whether the intervention is feasible with respect to participant recruitment rates, (iii) retention of pregnant women in the trial to 6 weeks postpartum; (iv) acceptability and feasibility of outcomes measures (to measure the efficacy within a definitive trial); (v) fidelity to the study protocol.

Secondary outcomes include: (i) Acceptability of the intervention. (ii) Process evaluation measures including rates of detection, referral and follow-up of high-risk pregnant women. (iii) Clinical outcomes of mean haemoglobin and mean systolic and diastolic blood pressures at 6 weeks postpartum.

Randomisation: Cluster randomisation will be conducted at the level of the PHC. Staff related to each PHC will be allocated to either intervention or control groups. The study will recruit 200 pregnant women across all 4 PHC clusters; 100 CHWs (known as ASHAs and ANMs) and; up to 8 Primary Care Physicians (affiliated to the PHC clusters). The villages selected under each intervention and control PHC will be non-contiguous to avoid contamination.

ELIGIBILITY:
Primary Health Centre cluster:

Inclusion Criteria:

* PHC serving population of greater than 30,000 people.
* Administrative lead for PHC consents for the PHC to participate in the study.

Exclusion Criteria:

* Administrative lead does not give consent for the PHC to participate in the study.

Pregnant women:

Inclusion Criteria:

* Age above 18 years.
* Participant is recruited between 28-36 weeks gestation.
* Participant is willing and able to give informed consent for participation in the study AND is:
* Living in the villages affiliated to the PHC included in the study.

Exclusion Criteria:

* Pregnant women who are younger than 18 years and;
* Pregnant women who are not recruited between 28-36 weeks' gestation
* Pregnant women not living in villages affiliated to the study PHCs will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 12 months
  Number of eligible pregnant women successfully recruited to study in 12 months.
Retention rate | 12 months
  Number of eligible participants who remain in study for entire duration up to and including the 6 week postpartum visit.
Number of home visits completed by Community Health Worker | 12 months
  Number of home visits completed by Community Health Worker using the SMARThealth Pregnancy mHealth platform in line with study protocol.

SECONDARY OUTCOMES:
Number of pregnant women diagnosed with gestational diabetes. | 12 months
  Number of participants correctly diagnosed with gestational diabetes mellitus using antenatal oral glucose tolerance test, in accordance with Government of India guidelines for Gestational Diabetes Mellitus, 2018.
Postpartum follow-up of pregnant women with gestational diabetes | 18 months
  Number of participants diagnosed with gestational diabetes who received postnatal 6 week oral glucose tolerance test, in accordance with Government of India guidelines for Gestational Diabetes Mellitus, 2018.
Number of pregnant women diagnosed with a hypertensive disorder of pregnancy. | 12 months
  Number of participants diagnosed with a hypertensive disorder of pregnancy using International Society for the Study of Hypertension in Pregnancy (ISSHP) criteria.
Number of pregnant women diagnosed with severe anaemia. | 12 months
  Number of participants diagnosed with severe anaemia (haemoglobin of <7g/dL) during pregnancy, in accordance with Government of India guidelines for Anaemia, 2018.
Mean postpartum haemoglobin | 12 months
  Haemoglobin values of postpartum women measured at 6 weeks postpartum.
Mean postpartum Systolic Blood Pressure | 12 months
  Systolic blood pressure of postpartum women measured at 6 weeks postpartum.
Mean postpartum Diastolic Blood Pressure | 12 months
  Diastolic blood pressure of postpartum women measured at 6 weeks postpartum.

CONTACTS AND LOCATIONS:
Locations (1):
- The George Institute for Global Health, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nagraj S, Kennedy S, Jha V, Norton R, Hinton L, Billot L, Rajan E, Mohammed Abdul A, Phalswal A, Arora V, Praveen D, Hirst J. A Mobile Clinical Decision Support System for High-Risk Pregnant Women in Rural India (SMARThealth Pregnancy): Pilot Cluster Randomized Controlled Trial. JMIR Form Res. 2023 Jul 20;7:e44362. doi: 10.2196/44362. PMID 37471135
- [Derived] Nagraj S, Kennedy SH, Jha V, Norton R, Hinton L, Billot L, Rajan E, Arora V, Praveen D, Hirst JE. SMARThealth Pregnancy: Feasibility and Acceptability of a Complex Intervention for High-Risk Pregnant Women in Rural India: Protocol for a Pilot Cluster Randomised Controlled Trial. Front Glob Womens Health. 2021 May 28;2:620759. doi: 10.3389/fgwh.2021.620759. eCollection 2021. PMID 34816187